CLINICAL TRIAL: NCT00727909
Title: Evaluation of Open-Ear Canal and Traditional Custom-Fit Hearing Aids
Brief Title: Evaluation of Open-canal Behind-the-Ear Hearing Aids and Traditional In-the-ear Hearing Aids.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C6288-R
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Hearing Loss
Keywords: Hearing loss; Hearing Aids; Speech Perception; Persons with Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hearing Aid Treatments (Experimental): Hearing aid treatments:
  TC (Traditional Custom), RITA (Receiver-in-the Aid), and RITE (Receiver-in the-Ear)
  Interventions: Device: Hearing Aid Treatments

INTERVENTIONS:
Device: Hearing Aid Treatments — Hearing aid treatments:
  Traditional Custom (TC), Receiver-in-the Aid (RITA) and Receiver-in-the-Ear (RITE)

SUMMARY:
This study is being conducted to evaluate the benefits of in-the-ear vs. open-fit behind-the-ear hearing aids. We want to learn more about which patients prefer each type, so we can make better choices about which type of hearing aid is best for which patients. Participants in this study will try three different sets of hearing aids for 2 months each, then we will evaluate the benefit of each type. Participants must be Veterans who are eligible for audiology care at one of the three participating sites.

DETAILED DESCRIPTION:
Hearing loss is the most common service-connected disability nationwide in the Veteran's Health Administration (VHA) system, with hearing aids providing the primary treatment option. Although the benefits of hearing-aid use are clearly established,~16-30% of adults who have hearing aids do not use them. Several factors are believed to result in non-use of traditional hearing aids, including (1) poor fit and comfort, (2) poor cosmetics, (3) whistling feedback, (4) occlusion, and (5) difficulty understanding speech in noise.

Recently, the open canal (OC) hearing-aid style has become a viable approach to addressing address many of the problems resulting in non-use of traditional hearing aids, particularly for individuals with mild to moderately-severe hearing loss. Although an OC hearing aid has many potential advantages, there also are potential limitations. For example, the maximum low and high-frequency gain available with an OC fitting is less than that available from traditional custom (TC) hearing-aid fittings, which could result in less than optimal amplification for some individuals. In addition, directional microphone benefits for speech understanding in noise, available with TC fittings, likely will be limited with OC fittings due to the loss of low-frequency gain (Ricketts et al., 2005).

Since both OC and TC fittings are appropriate for listeners with mild to moderately-severe hearing losses, evidence is needed to determine which style of hearing aid is preferred by a majority. Currently, OC fittings use a small behind-the-ear (BTE) hearing aid coupled to a thin tube or plastic covered wire ending in a vented "open" ear tip. When a TC fitting is used with patients with similar hearing losses, the majority are either an in-the-ear (ITE) or in-the-canal (ITC) .In the proposed study a comparison will be made between OC vs. TC fittings. In addition to this primary comparison, preference for one of two OC hearing aids, viz., OC instruments with receiver in the ear (OCRITE) and the OC instruments with receiver in the hearing-aid case (OCRIHA), will be determined. The outcomes of the OCRITE, OCRIHA, and TC hearing-aid use related to the factors of: (1) comfort and cosmetics, (2) subjective occlusion, (3) objective occlusion, (4) sound quality for external sounds, (5) feedback, (6) ease of use, (7) audibility, (8) aided signal-to-noise ratio (SNR) benefit, and (9) localization, will be measured in a large (n = 288), randomized-controlled, three-site (Bay Pines, Mountain Home, and Nashville) clinical trial, utilizing a three-period (two months each), cross-over design. A total of 13 variables will be measured for the 9 hearing-aid fitting and style-related factors. At the end of the study, participants will rank order their preferences for the three hearing aid fittings to determine (1) the preferred OC fitting (OCRITE vs. OCRIHA) and (2) whether the highest ranked OC fitting or the TC fitting is preferred. Preferred OC vs. TC difference scores will be calculated for all relevant variables. The ability of the differences scores to predict the preferences of the participants for an OC vs. TC hearing aid will be determined, in order to develop an evidence-based hearing aid selection model.

ELIGIBILITY:
Inclusion Criteria:

* Sensorineural hearing loss
* Veteran-adult onset of hearing
* English as first language
* Eligible for VA issued hearing aids
* Eligible to receive care at one of the three participating VA sites: Nashville, Tennessee, Mountain Home Tennessee, Bay Pines Florida

Exclusion Criteria:

* Known neurological, psychiatric disorders, or co-morbid disease that would prevent completion of the study
* Inadequate vision
* Inadequate reading skills

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2009-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gene W. Bratt, PhD MA BA, Principal Investigator — VA Medical Center
Locations (3):
- United States (3):
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - James H. Quillen VA Medical Center, Mountain Home, Tennessee
  - VA Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Veterans scheduled for audiology appointments at the three participating VA sites: Nashville, Tennessee, Bay Pines, Florida, and Mountain Home, Tennessee. Recruitment occurred during the time period May, 2009 through February, 2011.
Pre-assignment Details: All study participants were assigned into all three hearing aid treatments: Traditional Custom TC, Receiver-in-the Aid (RITA), Receiver-in-the-Ear (RITE). The sequence of treatments was counter-balanced to prevent an order effect.
  Eleven participants who consented withdrew or were excluded prior to the first condition hearing aid fitting.
Groups:
- TC RITE RITA: Participants received Traditional Custom hearing aid (TC) first, followed by Receiver in the Ear (RITE), followed by Receiver in the Aid (RITA). The length of each hearing aid treatment condition was 2 months.
- TC RITA RITE: Participants received Traditional Custom hearing aid (TC) first, followed by Receiver in the Aid (RITA), followed by Receiver in the Ear (RITE). The length of each hearing aid treatment condition was 2 months.
- RITE RITA TC: Participants received the Receiver in the Ear (RITE) hearing aid first, followed by Receiver in the Aid (RITA), followed by Traditional Custom hearing aid (TC). The length of each hearing aid treatment condition was 2 months.
- RITA RITE TC: Participants received the Receiver in the Aid (RITA) hearing aid first, followed by Receiver in the Ear (RITE), followed by Traditional Custom (TC). The length of each hearing aid treatment condition was 2 months.
Period: Overall Study
Arm/Group | TC RITE RITA | TC RITA RITE | RITE RITA TC | RITA RITE TC
Started | 65 | 72 | 67 | 75
Completed | 60 | 61 | 58 | 70
Not Completed | 5 | 11 | 9 | 5
Not completed — Withdrawal by Subject | 5 | 11 | 8 | 5
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Study Participants
Groups:
- All Study Participants: All study participants received all three hearing aid treatments (TC, RITA, RITE). The sequence of treatments was counter-balanced to prevent an order effect. Each hearing aid treatment lasted two months. Each treatment period was followed by the administration of a series of outcome measures before the next treatment was begun. At the conclusion of the third treatment, in addition to administration of the outcome measures, the participants were asked to rank the three hearing aid treatments in order of preference, and to provide subjective comments regarding the rationale for their rank-ordering.
Arm/Group | All Study Participants
Number analyzed (Participants) | 290
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 283
Region of Enrollment [Number; unit: participants]
  United States | 290

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Selected a Particular Type of Hearing Aid
Time Frame: At the end of the 6 month trial (after having worn each set of hearing aids for 2 months each)
Measure: Number; unit: percentage of participants
Groups:
- All Participants: All participants received all three hearing aid treatments.
Arm/Group | All Participants
Number analyzed (Participants) | 249
percentage of participants
  Percentage of participants preferring TC | 15
  Percentage of participants preferring RITE | 38
  Percentage of participants preferring RITA | 47

ADVERSE EVENTS:
Time Frame: 1 year, 10 months.
Description: The investigators at all 3 VA sites conducted their roles in this investigation under the purview of the local Institutional Review Board(IRB) at each site. The investigators, through their mandatory training, were fully cognizant of the significance of and procedures for reporting any adverse event that could have but did not occur.
Groups:
- All Study Participants: All participants received all three hearing aid treatments.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 1/290
Other Adverse Events (participants affected / at risk) | 0/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=290)
Congestive heart failure (Cardiac disorders) | 1 — Participant at Bay Pines died of congestive heart failure following hospitalization for hip fracture/hip surgery while enrolled in this study and in receipt of the second hearing aid intervention (RITA).The death was unrelated to study participation.

LIMITATIONS AND CAVEATS:
No limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No